CLINICAL TRIAL: NCT02090699
Title: Quantification of Diffuse Myocardial Iron Overload Related Interstitial Fibrosis With Cardiac Magnetic Resonance Imaging in Patients With Transfusion-Dependent Anemias
Brief Title: MR Imaging of Diffuse Myocardial Fibrosis in Transfusion-Dependent Anemias
Acronym: MAFIO
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Bernd Winterspersper, Dr. (MD), University Health Network, Toronto
Other Study IDs: RSNA-RR1318
Record Dates: First submitted 2014-02-28; First posted 2014-03-18 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Thalassemia Major; Chronic Blood Transfusion Related Iron Overload
Keywords: thalassemia major; chronic blood transfusion related iron overload; magnetic resonance imaging; myocardium; fibrosis
MeSH Terms: conditions — beta-Thalassemia; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myocardial Iron Overload: chronic blood transfusion related myocardial iron overload
- Healthy Volunteers: age matched healthy volunteers

SUMMARY:
Cardiac failure is the major cause of death in patients with thalassemia and chronic blood transfusion-related iron overload. The treatment of thalassemia has been revolutionized over the past decade with the implementation of cardiac MRI based assessment of iron overload. This has enabled detection of cardiac iron overload prior to symptomatic heart failure and now allows for timely therapy which has resulted in a substantial decrease in mortality. However, currently implemented MR imaging techniques assess for iron content only and not for iron related diffuse fibrosis which play a role in iron related heart failure. Histopathologic studies indicate that patients with iron overload have diffuse interstitial fibrosis. Quantitative MR techniques have shown that patients with various cardiomyopathies demonstrate diffuse myocardial fibrosis and that these changes correlate with changes in cardiac function. The investigators propose that quantitative cardiac MRI for assessment of diffuse myocardial fibrosis can further improve our ability to detect early damage to the myocardium and prevent morbidity and mortality from cardiac iron overload. Detection of fibrosis in patients with thalassemia may allow for earlier identification of cardiomyopathy when compared to other techniques in clinical use including T2* analysis. Identification of fibrosis could affect patient management as it would allow for tailoring of iron chelation therapy and may lead to better understanding of the disease processes contributing to heart failure and arrhythmia in these patients.

DETAILED DESCRIPTION:
Cardiac failure is the major cause of death in patients with transfusion-related iron overload. Histopathologic studies indicate that patients with myocardial siderosis have diffuse interstitial fibrosis. Cardiac MR assessment of the extracellular volume (ECV) fraction in other disease processes has been shown to accurately characterize diffuse myocardial fibrosis and to correlate with changes in diastolic function. No prior studies have assessed for diffuse interstitial myocardial fibrosis in patients with iron overload utilizing the proposed imaging techniques.

In this study, the investigators will assess the presence and extent of interstitial fibrosis in patients with transfusion-dependent anemias using cardiac MR techniques of T1 mapping and determination of ECV fraction. ECV values will be correlated with the severity of myocardial iron deposition determined by multi-echo T2*-weighted imaging, systolic ventricular function as determined by cardiac MR and diastolic function assessed by echocardiography. The investigators will recruit 35 patients with transfusion-related iron overload. Ten age-matched healthy subjects will be included as controls, to establish baseline values of myocardial T1 and ECV values. A modified Look-Locker with inversion recovery (MOLLI) sequence will be used to determine T1 values pre-, and post-administration of a gadolinium-based contrast agent (GBCA) at 1.5 Tesla. Calculated ECV values will be compared between iron-overload subjects and healthy controls, and will be correlated with left ventricular ejection fraction, measures of diastolic dysfunction and T2* values.

Detection of myocardial fibrosis in patients with iron overload would allow for improved prognostication and risk stratification. Elucidation of the relationship between myocardial fibrosis and myocardial iron deposition as well as cardiac functional parameters would provide valuable mechanistic insights and improved pathophysiological understanding of the disease. The results of the proposed study have the potential to significantly impact patient management including recommendations for earlier or more aggressive chelation therapy based on changes in ECV values.

ELIGIBILITY:
Inclusion Criteria (Patients):

Diagnosis of thalassemia Treatment with iron chelation therapy Referral for cardiac MR assessment of iron overload

Inclusion Criteria (Healthy Volunteers):

No significant past medical history and no evidence of cardiovascular or metabolic disease.

Exclusion Criteria (both groups):

Arrhythmia Claustrophobia Pregnancy and potential pregnancy (patient cannot exclude potential pregnancy) History of allergic reaction to Gadolinium based contrast agent (GBCA) Impaired renal function with eGFR < 30 ml/min/1.73m2 Any general MR contraindication such as pacemaker or defibrillators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with transfusion dependent anemias Age-matched healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evidence of diffuse myocardial fibrosis (elevated extracellular volume fraction) confirmed by MRI | at time of cardiac MR examination for each individual
  At the time of MRI respective imaging data will be collected to assess the extracellular volume fraction as a marker for diffuse myocardial fibrosis.

SECONDARY OUTCOMES:
Regional myocardial dysfunction as assessed by global longitudinal strain Echocardiography measurement | at time of echocardiography examination for each individual
  At the time of echocardiography (same day as MRI) respective strain data with be gathered for outcome assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hanneman K, Nguyen ET, Thavendiranathan P, Ward R, Greiser A, Jolly MP, Butany J, Yang IY, Sussman MS, Wintersperger BJ. Quantification of Myocardial Extracellular Volume Fraction with Cardiac MR Imaging in Thalassemia Major. Radiology. 2016 Jun;279(3):720-30. doi: 10.1148/radiol.2015150341. Epub 2015 Dec 10. PMID 26653680